CLINICAL TRIAL: NCT06287489
Title: Effects of Mediterranean Diet on Physical and Cognitive Functions in Community-dwelling Older People With Subjective Cognitive Decline - a Randomized Controlled Cross-over Trial
Brief Title: Effects of Mediterranean Diet on Subjective Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chih-Ping Chung (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor-Investigator, Chih-Ping Chung, Professor M.D., Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: No.:2023-08-010ACF
Record Dates: First submitted 2024-02-16; First posted 2024-03-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Subjective Cognitive Decline
MeSH Terms: interventions — Diet, Mediterranean; Diet

STUDY DESIGN:
Intervention Model Description: Mediterranean diet phase X regular diet phase
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet phase followed by regular diet phase (Other): Three-month of M phase, one month of washout and three month of R phase
  Interventions: Other: Mediterranean diet; Other: Regular diet
- Regular diet phase followed by Mediterranean diet phase (Other): Three-month of R phase followed by three month of M phase
  Interventions: Other: Mediterranean diet; Other: Regular diet

INTERVENTIONS:
Other: Mediterranean diet — Mediterranean diet for three month
Other: Regular diet — regular diet

SUMMARY:
Research Questions:

1. Due to the fact that most participants in past clinical trials on the Mediterranean diet were cognitively healthy individuals, and while the observed effects were significant, they were not particularly substantial, does the Mediterranean diet have similarly significant and more pronounced effects on both physical and cognitive functions in older adults with subjective cognitive decline (SCD)?
2. What is the mechanism behind the effects of the Mediterranean diet on physical or/and cognitive function? Is it through vascular protection or improvements in brain structure/brain network function?

Research Objective:

Conduct a cross-over randomized controlled trial to investigate the effects of a three-month Mediterranean diet on the physical and cognitive functions of older adults with subjective cognitive decline (SCD) in the community. Utilize brain MRI and circulatory biomarkers measurements to elucidate the underlying mechanisms.

DETAILED DESCRIPTION:
Research Questions:

1. Due to the fact that most participants in past clinical trials on the Mediterranean diet were cognitively healthy individuals, and while the observed effects were significant, they were not particularly substantial, does the Mediterranean diet have similarly significant and more pronounced effects on both physical and cognitive functions in older adults with subjective cognitive decline (SCD)?
2. What is the mechanism behind the effects of the Mediterranean diet on physical or/and cognitive function? Is it through vascular protection or improvements in brain structure/brain network function?

Research Objective:

Conduct a randomized controlled trial to investigate the effects of a three-month Mediterranean diet on the physical and cognitive functions of older adults with subjective cognitive decline (SCD) in the community. Utilize brain MRI to elucidate the underlying mechanisms.

Participants inclusion criteria:

SCD-plus subjects must fullfill the following five criteria

1. Subjective memory decline without impairment in other cognitive domains (MMSE > 26; MMSE > 14 for those with less than six years of education).
2. Onset of subjective cognitive decline within the past 5 years.
3. Age at the onset of subjective cognitive decline is greater than 60 years.
4. Concern and preoccupation with the decline in memory.
5. Perceived functional decline relative to peers and meet one of the following three criteria:

   1. Caregiver perceives cognitive decline.
   2. Carries the APOE ε4 genotype.
   3. Clinical evidence of preclinical Alzheimer's disease biomarkers.

Participants exclusion criteria:

1. Cases unable to comply with or accept the dietary intervention, including individuals with dietary restrictions such as vegetarianism, lactose intolerance, or potential food allergies.
2. Walking speed ≤ 0.3 meters/second.
3. Any significant medical conditions affecting physical and cognitive functions, including:

   1. Limb fracture within the past six months.
   2. Severe arthritis within the past six months.
   3. Neurological and psychiatric disorders as determined by the principal investigator (e.g., stroke, Parkinson's disease, peripheral neuropathy, mental disorders).
   4. Intermittent claudication due to peripheral arterial disease.
4. Chronic kidney disease (eGFR <30 ml/min/1.73m2) and individuals undergoing dialysis.
5. Poorly controlled cardiovascular diseases as determined by the principal investigator.
6. Poorly controlled malignant tumors as determined by the principal investigator.
7. Severe visual and hearing impairments preventing the completion of assessments and tests.
8. Participants who have undergone hormone therapy in the three months preceding the trial or are expected to undergo hormone therapy during the trial.

Study Design or Implementation:

This study is a cross-over (three month of Mediterranean diet phase "M" and three month of regular diet phase "R") randomized controlled trial with a duration of six to seven months (seven month for MR group with an additional one-month washout period). During the study period, participants in the M phase will receive a daily portion of a Mediterranean diet designed by a nutritionist. Regular Mediterranean diet education and reviews will be conducted to ensure that the Mediterranean Diet Score System (MDSS) reaches a score of ≥10. The R phase will follow a self-selected diet, and the MDSS during then will also be assessed.

Eligible participants will be randomly assigned to two groups with different diet sequences (MR or RM group) in a 1:1 ratio. T0 measurements will be conducted, including a basic information questionnaire, blood biomarker sampling for Alzheimer's disease, and the initial assessment of physical and cognitive functions. Dietary assessments and education will be conducted before entering the dietary intervention group and at one week, two weeks, one month, two months, and three months after entering each phase. Other measurements, including blood pressure, heart rate, height and weight measurements, blood tests, and brain MRI, will be performed at T1 and T2 (end of each diet phase).

ELIGIBILITY:
Inclusion Criteria:

Subjective cognitive decline (SCD)-plus subjects, individuals must meet five criteria:

1. Subjective memory decline without impairment in other cognitive domains (MMSE > 26; MMSE > 14 for <6 years of education).
2. Onset of subjective cognitive decline within the past 5 years.
3. Age at the onset of subjective cognitive decline is >60 years.
4. Concern and preoccupation with memory decline.
5. Perceived functional decline relative to peers and meet one of three criteria: a. Caregiver perceives cognitive decline; b. Carries APOE ε4 genotype; c. Clinical evidence of preclinical Alzheimer's disease biomarkers.

Exclusion Criteria:

Exclude individuals who:

1. Cannot comply with or accept the dietary intervention (e.g., dietary restrictions, vegetarianism, lactose intolerance).
2. Have walking speed ≤ 0.3 meters/second.
3. Have significant medical conditions affecting physical and cognitive functions.
4. Have chronic kidney disease (eGFR <30 ml/min/1.73m2) or undergo dialysis.
5. Experience poorly controlled cardiovascular diseases or malignant tumors.
6. Have severe visual and hearing impairments preventing assessments.
7. Have undergone hormone therapy in the preceding three months or are expected to during the trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Cognitive functional change | Three month of allocated diet phase
  Subjective and objective cognitive functional measurements (MMSE and comprehensive neuropsychological tests for verbal memory, attention, visuospatial function, executive function, and language)
Physical function 1 - gait speed change | Three month of allocated diet phase
  Gait speed measurements
Physical function 2 - handgrip strength change | Three month of allocated diet phase
  Handgrip strength measurements
Physical function 3 - stand from chair speed change | Three month of allocated diet phase
  Five times of stand from chair speed measurements
Brain MRI structural change - total and regional voxel-based brain parenchymal features change | Three month of allocated diet phase
  Brain gray matter/white matter volumes and diffusion tensor imaging measurements
Brain MRI functional change - total and regional voxel-based brain functional features change | Three month of allocated diet phase
  Resting functional MRI signal analsyes
Brain MRI neurovascular lesion change - small vessel disease markers | Three month of allocated diet phase
  white matter hyperintensities, lacune and cerebral microbleeds assessments
Brain MRI neurovascular structural change - microvascular density | Three month of allocated diet phase
  arteriolar and venular densities

SECONDARY OUTCOMES:
AD circulatory biomarkers | Three month of allocated diet phase
  Amyloid beta 40/42, p-tau-217, NfL, TDP43,ASC level changes

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ping Chung, MD PhD, Principal Investigator — Department of Neurology, Neurological Institute, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No